CLINICAL TRIAL: NCT02009501
Title: A Prospective, Open, Comparative, Randomized Single-center Study to Evaluate the Effect of V.A.C. VeraFlo™ Therapy With .125% Dakins vs V.A.C. Ulta™ Therapy on Biofilm Removal/Disruption/Elimination in Chronically Infected Wounds
Brief Title: V.A.C. VeraFlo™ Instillation Therapy vs V.A.C. Ulta™ Therapy on Biofilm in Chronically Infected Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: Kinetic Concepts, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAC/09/05/ULTA
Record Dates: First submitted 2013-11-24; First posted 2013-12-12 (Estimated); Results first posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Lower Extremity Wound Infected; Venous Stasis Ulcers
Keywords: Infected wounds; NPWTi; VAC Instill; Biofilm
MeSH Terms: conditions — Varicose Ulcer; Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VAC VeraFlo with Dakins Instillation (Active Comparator): VAC VeraFlo with Dakins .125% instillation will be initially applied in the OR after surgical debridement. Dressing will be changed on day 4 and and removed on day 7. Wound assessments will continue at weeks 2, 3, and 4.
  Interventions: Device: VAC VeraFlo with Dakins Instillation
- VAC Ulta Therapy (Active Comparator): VAC ULTA Therapy will be initially applied in the OR after surgical debridement. Dressing will be changed on day 4 and and removed on day 7. Wound assessments will continue at weeks 2, 3, and 4.
  Interventions: Device: VAC Ulta Therapy

INTERVENTIONS:
Device: VAC VeraFlo with Dakins Instillation — VAC VeraFlo with Dakins instillation will be placed in the operating room after surgical debridement. Biopsies will be obtained prior to surgical debridement, after surgical debridement, on day 4, and on day 7.
  Other Names: NPWTi; VAC Instill
  Arms: VAC VeraFlo with Dakins Instillation
Device: VAC Ulta Therapy — VAC ULTA will be placed in the operating room after surgical debridement. Biopsies will be obtained prior to surgical debridement, after surgical debridement, on day 4, and on day 7.
  Other Names: VAC; NPWT
  Arms: VAC Ulta Therapy

SUMMARY:
This study would like to determine if using negative pressure wound therapy with an instillation of .125% Dakins is more effective than using negative pressure wound therapy alone on biofilm removal, disruption and elimination in chronically infected lower extremity wounds.

ELIGIBILITY:
Inclusion Criteria:

* The patient is of 18 years or older.
* Males and females - provided they are not pregnant and if of reproductive age are using contraception.
* Patient with ulcers that:

  1. Have an ulcer area of at least 4 cm2 confirmed via counting squares on an wound tracing
  2. Have been present for at least 4 weeks
  3. Are confirmed to have a colony forming unit per gram of wound tissue greater than or equal to 10 to the 5th cfu
  4. Are full thicknesses through to dermal or subcutaneous tissue but not extending to muscle or bone.
  5. The patient has an ABI of greater or equal to 0.8 and lower than 1.3 or has a suitable Peripheral Vascular Resistance (PVR) and Doppler assessment which confirms venous disease & therefore treatment with Profore is deemed acceptable by the clinician.
  6. The patient has one or more clinical signs of infection (edema, malodor, local/periwound erythema, spontaneous pain between dressing changes, increased exudate, discoloration of granulation tissue, increased temperature at wound, non progression of wound, purulent exudate and friable granulation tissue)
  7. The patient is able to understand the evaluation and is willing to consent to the evaluation.
  8. Patients with a suitable wound on a different limb to any other wounds previously eligible.

Exclusion Criteria:

1. Patients undergoing chemotherapy
2. Patients being treated with immunosuppressive drugs or corticosteroids
3. Patients with an autoimmune disease
4. Patients who have participated in an experimental drug or device study within the last 15 days
5. Patients that have been entered in this evaluation previously as an evaluable patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C Lantis, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- St. Luke's-Roosevelt Hospital Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began Nov 2013, with enrollment in Jan 2014 and trial conducted to Nov 2014. All patients were recruited from the outpatient vascular and wound care clinic at Mt Sinai St Luke's - Roosevelt Hospitals in New York City.
Groups:
- VAC Ulta Therapy: VAC ULTA Therapy applied in the OR after surgical debridement.
- VAC VeraFlo With Dakins Instillation: VAC VeraFlo with Dakins Instillation.0.125% instillation applied in the OR after surgical debridement.
Period: Overall Study
Arm/Group | VAC Ulta Therapy | VAC VeraFlo With Dakins Instillation
Started | 9 | 11
Completed | 9 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VAC Ulta Therapy | VAC VeraFlo With Dakins Instillation | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (2.4) | 62.3 (5.8) | 63.83 (4.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 7 | 9 | 16
Ulcer duration [Mean (Standard Deviation); unit: months] | 93.9 (42.9) | 103.3 (43.3) | 99.07 (43.37)
Ulcer size [Mean (Standard Deviation); unit: cm^3] | 43.5 (10.8) | 56.2 (17.8) | 50.48 (16.33)
Etiology [Count of Participants; unit: Participants]
  Venous | 5 | 7 | 12
  Diabetic | 0 | 1 | 1
  Mixed | 4 | 3 | 7
Comorbidities [Count of Participants; unit: Participants]
  Hypertension | 6 | 7 | 13
  Diabetes Mellitus | 6 | 5 | 11
  Morbid Obesity | 1 | 2 | 3
  Chronic Kidney Disease | 1 | 2 | 3
  Hyperlipidemia | 6 | 7 | 13
  Tobacco use | 3 | 7 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Bacteria Colony-forming Units Using When NPWT and NPWTi on Venous Leg Ulcers
Description: Biopsies for bacteria colony-forming units obtained at pre surgical debridement (baseline) and day 7.
Time Frame: Baseline and day 7
Measure: Mean (Standard Deviation); unit: 10^3 CFU/g
Arm/Group | VAC Ulta Therapy | VAC VeraFlo With Dakins Instillation
Number analyzed (Participants) | 9 | 11
10^3 CFU/g
  Baseline | 8.6 (8.8) | 12.9 (12.5)
  7 days post application | 2.5 (5.0) | 3.2 (9.4)

ADVERSE EVENTS:
Description: Adverse events not collected
Arm/Group | VAC Ulta Therapy | VAC VeraFlo With Dakins Instillation
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Limitation: small sample size and associated large data variance. Absence of a standardized biopsy schema given the heterogeneous distribution of biofilm-protected bacteria within wounds, may not properly capture effects of the treatment modalities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes